CLINICAL TRIAL: NCT00463983
Title: Phase 2 Study of Long Acting Octreotide in Idiopathic Pulmonary Fibrosis
Brief Title: Treatment of Idiopathic Pulmonary Fibrosis with Long Acting Octreotide
Acronym: FIBROSAND
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: C05-32
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- octreotide (Experimental): octreotide SR 30 mg intra muscularly every 4 weeks
  Interventions: Drug: octreotide

INTERVENTIONS:
Drug: octreotide

SUMMARY:
Octreotide is a somatostatin analog with a long half-life in vivo. Octreotide has interesting anti-inflammatory and anti-fibrotic properties in vitro and in vivo. Somatostatin receptors are increased and Octreotide uptake is increased in the lung in patients with idiopathic pulmonary fibrosis. Our hypothesis is that octreotide may slow the degradation of lung function in patients with IPF. In this proof of concept study, patients with IPF will receive an intramuscular injection of slow release octreotide (Sandostatin LP, 30 mg)every 4 weeks for 48 weeks. Lung function (FVC, DLCO), HRCT scores for fibrosis and ground glass, 6 minute walking test,quality of life and survival will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* confident diagnosis of IPF according to ATS/ERS criteria

Exclusion Criteria:

* known intolerance to somatostatin or octreotide
* another disease with predicted survival < 12 months
* pregnancy or lactation
* previous treatment with somatostatin or somatostatin analogs
* patient on a waiting list for transplantation
* antifibrotic treatment or prednisone > 10 mg/day within the last 6 weeks
* symptomatic biliary lithiasis
* blood coagulation disorders that prevent intra-muscular injections
* HIV infection
* hepatitis B or C active infection

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-10; Primary Completion 2010-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
FVC changes | 12 months

SECONDARY OUTCOMES:
DLCO changes | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Crestani, MD, PhD, Principal Investigator — INSERM, France
Locations (16):
- France (16):
  - Service de Pneumologie Hôpital Avicenne 125 rue de Stalingrad, Bobigny
  - Service de Pneumologie Hôpital Ambroise Paré, Boulogne-Billancourt
  - Service de Pneumologie Hôpital Côte de Nacre, Caen
  - Service de Pneumologie Hôpital Antoine Béclère, Clamart
  - Service de Pneumologie Centre hospitalier intercommunal de Créteil, Créteil
  - Service de Pneumologie Hôpital Albert calmette, Lille
  - Service de Pneumologie Hôpital Sainte Marguerite BP 29, Marseille
  - Service de Pneumologie Hôpital Saint-Antoine, Paris
  - Hôpital Bichat 46 rue Henri Huchard, Paris
  - Service de Pneumologie A Hôpital Bichat 1, Paris
  - Service de Pneumologie Hôpital Saint Louis 1 avenue Claude-Vellefaux, Paris
  - Service de Pneumologie Hôpital de la Pitié-Salpetrière 47-83 boulevard de l'hôpital, Paris
  - Service de Pneumologie Hôpital Cochin, Paris
  - Service de Pneumologie Hôpital Georges Pompidou, Paris
  - Service de Pneumologie A Hôpital Tenon, Paris
  - Service de Pneumologie Hôpital Pontchaillou, Rennes

REFERENCES:
- [Background] Crestani B, Chapron J, Wallaert B, Bergot E, Delaval P, Israel-Biet D, Lacronique J, Monnet I, Reynaud-Gaubert M, Tazi A, Lebtahi R, Debray MP, Brauner M, Dehoux M, Dornic Q, Aubier M, Mentre F, Duval X. Octreotide treatment of idiopathic pulmonary fibrosis: a proof-of-concept study. Eur Respir J. 2012 Mar;39(3):772-5. doi: 10.1183/09031936.00113011. No abstract available. PMID 22379151
- [Background] Lebtahi R, Moreau S, Marchand-Adam S, Debray MP, Brauner M, Soler P, Marchal J, Raguin O, Gruaz-Guyon A, Reubi JC, Le Guludec D, Crestani B. Increased uptake of 111In-octreotide in idiopathic pulmonary fibrosis. J Nucl Med. 2006 Aug;47(8):1281-7. PMID 16883006